





**Full Title** The African Critical Illness Outcomes Study

Short Title ACIOS

**Sponsor** Department of Anaesthesia and Perioperative Medicine, University of Cape

Town, Anzio Road, Cape Town 7925

Funder National Institute for Healthcare and Care Research (NIHR) through the

Global Health Group on Perioperative and Critical Care: "APPRISE"

**Chief Investigator** Tim Baker

Department of Emergency Medicine

Muhimbili University of Health and Allied Sciences

Dar es Salaam

Tanzania

Email: tim.baker@ki.se

Telephone: +255 68 323 6765

**Co-Chief Investigators** Bruce Biccard

Department of Anaesthesia and Perioperative Medicine

University of Cape Town

South Africa

Email: <a href="mailto:bruce.biccard@uct.ac.za">bruce.biccard@uct.ac.za</a>
Telephone: +27 (0) 76 160 6387

**Rupert Pearse** 

Professor & Consultant in Intensive Care Medicine

Queen Mary University of London and Barts Health NHS Trust

Royal London Hospital

London

**United Kingdom** 

Email: <u>r.pearse@qmul.ac.uk</u> Tel: +44 (0)20 3594 0351

Statistician Anneli Hardy

NIHR Global Health Group on Perioperative and Critical Care: "APPRISE"

**Data management** Safe Surgery South Africa








# 1. Signature page

#### **CI Agreement**

The study, as detailed within this Research Protocol, will be conducted in accordance with the principles of GCP, and the Declaration of Helsinki (64th WMA General Assembly, Fortaleza, Brazil, October 2013) and any other applicable regulations. I delegate responsibility for the statistical analysis and oversight to a qualified statistician (see declaration below).

CI name: Tim Baker

Signature:

Date: 17 April 2023

Tim Baker

#### Statistician's Agreement

The study as detailed within this research protocol will be conducted in accordance with the World Medical Association Declaration of Helsinki (64th WMA General Assembly, Fortaleza, Brazil, October 2013), Principles of ICH E6-GCP, ICH E9 - Statistical principles for Clinical Trials and ICH E10 - Choice of Control Groups.

I take responsibility for the statistical work in this protocol is accurate and take responsibility for statistical analysis and oversight in this study.

Statistician's name: Anneli Hardy

Signature:

Date: 17 April 2023







# **Contents**

| 1. | Sign | ature page | 2 |
|----|---------|-----------------------------------------------|------|
| 2. | List | of abbreviations | 5 |
| 3. | Sum | mary | 6 |
| 4. | Intro | oduction | 7 |
| 5. | Aim | , Objectives, Research questions and Outcomes | 8 |
| | 5.1 | Aim | 8 |
| | 5.2 | Objectives | 8 |
| | 5.3 | Research questions | 8 |
| | 5.4 | Co-primary outcomes | 9 |
| | 5.5 | Secondary outcomes | 9 |
| | 5.6 | Hospital level outcome | 9 |
| 6. | Met | hods | 9 |
| | 6.1 | Study design | 9 |
| | 6.2 | Study setting | 9 |
| | 6.3 | Hospital participation criteria | 9 |
| | 6.4 | Study population (patient Inclusion criteria) | 9 |
| | 6.5 | Exclusion criteria | 9 |
| 7. | Stuc | ly Procedures | . 10 |
| | 7.1 | Hospital Recruitment | . 10 |
| | 7.2 | Study data | . 10 |
| | 7.3 | Data collection | . 10 |
| | 7.3. | 1 Schedule of assessment | . 10 |
| | 7.3. | 2 Hospital level data collection | . 10 |
| | 7.3. | 3 Patient level data collection | . 11 |
| | 7.3. | 4 Outcomes | . 11 |
| | 7.4 | End of Study Definition | . 12 |
| 8. | Defi | nitions | . 12 |
| 9. | Data | a Handling and Management | . 13 |
| 10 | . Stat | istical Analysis | . 14 |
| | 10.1 S | ample size calculation | . 14 |
| | 10.2 St | atistical analysis | . 14 |
| 11 | Ethi | cal Considerations | . 15 |







| 12. | Safety considerations | 16 |
|-----|------------------------------------|----|
| 13. | Monitoring and Auditing | 16 |
| 14. | Study Committees | 16 |
| 1 | 4.1 Study Management Team | 16 |
| 1 | 4.2 Steering Committee | 17 |
| 1 | 4.3 Country Coordinators | 17 |
| 1 | 4.3 Local Coordinators | 17 |
| 15. | Dissemination and Publication Plan | 17 |
| 16. | Deliverables | 18 |
| 17. | Finance and Funding | 18 |
| 18. | References | 18 |
| Δnn | endices | 21 |







# 2. List of abbreviations

ACCCOS African COVID-19 Critical Care Outcomes Study

ACIOS African Critical Illness Outcomes Study

APORG (African Perioperative Research Group)

APPRISE African Partnership on Perioperative and Critical Care Research

ASOS African Surgical Outcomes Study

ASOS-2 African Surgical OutcomeS-2 (ASOS-2) trial

CRISPOS Critical Illness and Sepsis Prevalence and Outcomes Study

EECC Essential Emergency and Critical Care

EuSOS European Surgical Outcomes Study

HDU High Dependency Unit

ICU Intensive Care Unit

ISOS International Surgical Outcomes Study

NIHR National Institute for Health and Care Research

SAP Statistical Analysis Plan







# 3. Summary

| Short title | ACIOS |
|---|---|
| Methodology | A prospective, international, multi-centre, observational study. |
| Research sites | Acute hospitals in African countries. |
| Objective | To determine the hospital point-prevalence and mortality rates of |
| | adult patients with critical illness in hospitals in Africa. |
| Number of patients | Not specified. All eligible patients in participating hospitals. |
| Inclusion criteria | All in-hospital patients aged 18 years or older in all departments and |
| | wards in participating hospitals in Africa. |
| Exclusion criteria | None |
| Patient follow-up | Until hospital discharge or death, censored at 7 days after inclusion. |
| Primary | 1. The presence of critical illness |
| outcomes | 2. 7-day in-hospital mortality |
| Statistical | Descriptive statistics, univariate and multivariable logistic regression |
| analysis | models. A statistical analysis plan will be written before analysis. |
| Data collection | One day in each hospital in September-November 2023 plus 7 days |
| duration | follow-up in each hospital |
| Proposed start | 1 <sup>st</sup> September 2023 |
| date | |
| Proposed end | 7 <sup>th</sup> December 2023 |
| date | |







#### 4. Introduction

Critically ill patients – those in *a state of ill health with vital organ dysfunction, a high risk of imminent death if care is not provided, and the potential for reversibility*.¹ – have particular needs, and managing these needs is a core function of hospitals. Triage at admission and on the wards is needed to identify these patients with critical illness.²,³ Critically ill patients need regular contact with health workers and close observation and frequent modifications to care, either in general wards, or in specialised locations such as Intensive Care Units (ICUs) and High Dependency Units (HDUs).⁴ Rapid Response Teams of acute care specialists may be implemented in hospitals to provide care when called by ward staff.⁵

There are reports of gaps in the readiness and provision of critical care in hospitals in Africa.<sup>6-8</sup> Essential Emergency and Critical Care (EECC) has been developed and defined as the first-line care that should be provided to all critically ill patients.<sup>9,10</sup> Focusing on the first-line care in EECC is a strategy to address the gap in critical care. In our previous work an unmet need of EECC of 50-90% was found in hospitals in Malawi,<sup>8</sup> and there have been many calls to increase the coverage of EECC to address this gap.<sup>9,11-13</sup>

While it is accepted that critical illness and the underlying causes of critical illness are common, the number of patients with critical illness has not been accurately quantified. In one region of Sweden we found 10% of hospital inpatients to be critically ill, and in a Tanzanian university hospital's emergency unit, 10% of patients were critically ill at arrival. Global estimates have been attempted by using the admission rates to ICUs but this method reflects national and local uses of ICUs which vary greatly even between high-income countries. The indirect annual global estimate of 30-45 million adults made by extrapolating the incidence of common diseases leading to critical illness in North America is likely to be an underestimate as the burden of disease is greater in settings of lower resources. Moreover, the mortality of critically ill patients has not been accurately quantified, with reports of 18-82% in-hospital mortality rates. The indirect annual global estimate of 30-45 million adults made by extrapolating the incidence of common diseases leading to critical illness in North America is likely to be an underestimate as the burden of disease is greater in settings of lower resources. Moreover, the mortality of critically ill patients has not been accurately quantified, with reports of 18-82% in-hospital mortality rates.

A patient's vital signs (heart rate, respiratory rate, blood pressure, conscious level, body temperature, oxygen saturation) are commonly used measurements in hospital care. Deranged vital signs have been shown to correlate with negative outcomes such as admission to the ICU,<sup>26,27</sup> unexpected cardiac arrest,<sup>27,28</sup> and mortality,<sup>27,29</sup> and are pragmatic and useful as criteria for the identification of critical illness.<sup>30,31</sup>







We will conduct a prospective, international, multi-centre, observational study of all adult in-patients in hospitals across Africa, based on the methods we developed in the International Surgical Outcomes Study (ISOS),<sup>32</sup> European Surgical Outcomes Study (EuSOS),<sup>33</sup> African Surgical Outcomes Study (ASOS),<sup>34</sup> and African COVID-19 Critical Care Outcomes Study (ACCCOS)<sup>22</sup> studies. Using vital-signs based criteria, we will determine the hospital point-prevalence of critical illness. We will collect data on the care provided to patients, so to determine the coverage of essential emergency and critical care. We will follow the adult in-hospital patients for 7 days or until hospital discharge (whichever is sooner), allowing an estimate of the mortality rate and patients at increased risk who are critically ill in this population. The knowledge generated in the ACIOS study will assist in improving organisation of acute hospital services with the goal of averting substantial numbers of preventable deaths in African hospitals.

# 5. Aim, Objectives, Research questions and Outcomes

#### 5.1 Aim

To investigate critical illness, its care and associated outcomes among all adult inpatients in hospitals across Africa.

#### 5.2 Objectives

- 1. To establish the proportion of adult (18 years or older) inpatients in African hospitals that are critically ill.
- 2. To establish the mortality rate of the critically ill patients and those who are not critically ill.
- 3. To estimate the proportion of critically ill patients who receive essential emergency and critical care.
- 4. To investigate the association between the provision of essential emergency and critical care to critically ill patients and mortality.
- 5. To determine the availability of resources for essential emergency and critical in African hospitals.

#### 5.3 Research questions

Among adult (18 years or older) inpatients in African hospitals:

- 1. What proportion of patients are critically ill?
- 2. What are the mortality rates for patients who are, and who are not critically ill?
- 3. What proportion of critically ill patients receive essential emergency and critical care?
- 4. What is the relationship between essential emergency and critical care provision, and mortality? In African hospitals:








5. What is the availability of resources for the provision of essential emergency and critical care?

## 5.4 Co-primary outcomes

- Presence of critical illness
- In-hospital mortality (censored at 7-days)

## 5.5 Secondary outcomes

- Provision of essential emergency and critical care
- Length of hospital stay

### 5.6 Hospital level outcome

Availability of resources for essential emergency and critical care

#### 6. Methods

# 6.1 Study design

African, multi-centre prospective observational cohort study of in-hospital adult patients.

# 6.2 Study setting

Hospitals across Africa.

# 6.3 Hospital participation criteria

Any acute hospital in Africa providing adult inpatient care (see Definitions section 8).

# 6.4 Study population (patient Inclusion criteria)

All adult patients aged 18 years or over who have been admitted for inpatient care in any department or ward in participating hospitals.

#### 6.5 Exclusion criteria

None.







# 7. Study Procedures

## 7.1 Hospital Recruitment

Hospitals will be recruited through the African Perioperative Research Group (APORG) network, the Essential Emergency and Critical Care (EECC) network and other networks in Africa.

#### 7.2 Study data

Data will be collected on all eligible patients on the study day and then during in-hospital follow-up.

#### 7.3 Data collection

A pragmatic and realistic dataset is fundamental to the success of the study. Data will be collected on paper on one-day in each hospital plus follow-up censored at 7 days. Data will be collected:

- At hospital level for the availability of resources for EECC.
- At the patient's bedside for patient demographic and medical information, physiological signs,
   and ongoing provision of EECC and
- From hospital records for patient outcomes.

#### 7.3.1 Schedule of assessment

| Event/ Visit | Study day | Until discharge or death, censored at 7 days |
|---|---|---|
| Hospital level data | X | |
| Inclusion/ exclusion criteria | X | |
| Demographic information | Х | |
| Medical information | X | |
| Physiological signs | X | |
| EECC provision | X | |
| Outcomes | | X |

# 7.3.2 Hospital level data collection

Data will be collected once for each hospital to assess the availability of resources for the provision of EECC. A checklist of resources will be used and data entered together with a key informant in the hospital. The key informant may be the medical-officer-in-charge or other clinician or administrator







who has an in-depth knowledge of the resources available in the hospital for managing critically ill patients, as identified by the study team's local coordinator. In addition, data will be collected on:

- Population served (catchment area)
- Primary, secondary or tertiary hospital
- Number of hospital beds
- Number and level of critical care beds
- Details about the reimbursement status of the hospital
- Resources in the hospital such as staff and equipment

#### 7.3.3 Patient level data collection

On the specified day of data collection, every patient fulfilling the inclusion criteria in every department and ward in the hospital will be included in the study. Patients who are absent from their beds when the study team arrive, (for example, are in an operating theatre, or undergoing a medical investigation), will be re-visited later the same day and included when they are back in their bed, or when they are in a bed where inclusion is possible such as in a surgical recovery room. Data on patient demographics, medical information and current care provided will be collected from the patient and from the clinical team. The patient's vital sign measurements, (respiratory rate, oxygen saturation, blood pressure, heart rate, conscious level), will be checked by the study team using the hospital's equipment. If it is inappropriate for a patient's vital signs to be checked – for example if the clinical team has made the decision to refrain from vital sign observations as the patient is in the final stage of dying, (may be termed 'on an end-of-life pathway', "moribund", 'gasping' or 'late palliative phase' by the clinical team), or if the patient refuses permission to measure their vital signs – then the patient will be included in the study but vital signs will not be measured. It will be acceptable for the study team to record the last vital signs recorded in the patient's file for these patients. For women in active labour, the vital signs will be measured between contractions. Detailed data collection procedures will be described in the study's Standard Operating Procedures. Data will be collected by clinician investigators, and/ or clinician researchers working at the site.

#### 7.3.4 Outcomes

The patient outcomes will be reported as alive and discharged, died, or alive and still in hospital censored at 7-days.








### 7.4 End of Study Definition

The end of the study is defined as the end of the 7-day follow-up for the last included patient. Data analysis shall follow this.

#### 8. Definitions

*Critical illness (co-primary outcome):* a state of ill health with vital organ dysfunction, a high risk of imminent death if care is not provided and the potential for reversibility. Patients will be classified as critically ill if they have one or more severely deranged vital signs as in Figure 1. The cut-offs are those used in the Critical Illness and Sepsis Prevalence and Outcomes Study (CRISPOS) study and based on previous research in Tanzania and Sweden<sup>30,35,36</sup>:

| Criterion | Vital signs | Definition critically ill |
|-----------------|--------------------------------|---------------------------|
| Conscious level | Conscious level (AVPU Scale) | P or U |
| Respiratory | Respiratory rate per minute | <8 or >30 |
| | Oxygen saturation (%) | <90 |
| Circulatory | Heart rate per minute | <40 or >130 |
| | Systolic blood pressure (mmHg) | <90 |

Figure 1: Criteria for the definition of critical illness

*Hospital population:* all adult patients aged 18 years or over who have been admitted for inpatient care in any department or ward in participating hospitals on the day of data collection.

Essential Emergency and Critical Care (EECC): the care that all critically ill patients should receive, in all hospitals in the world including clinical processes such as oxygen therapy, intravenous fluids and patient positioning to protect the airway, as described in the 2021 global consensus.<sup>10</sup>

*Availability of resources for EECC*: The 66 resources necessary for the provision of EECC including items such as pulse oximeters, oxygen masks and intravenous fluids.<sup>10</sup>

*Coverage of EECC*: The proportion of critically ill patients receiving EECC.

Patients will be deemed to be receiving EECC if they are:

- critically ill due to the conscious level criterion (Figure 1) <u>and</u>:
  - o are lying in the lateral position **or**







- o have an oro-pharyngeal or naso-pharyngeal airway inserted in their pharynx <u>or</u>
- o have an ongoing chin-life or jaw-thrust or
- o have other airway protection
- critically ill due to a respiratory criterion (Figure 1) <u>and</u>:
  - o are receiving oxygen
- critically ill due to a circulatory criterion (Figure 1) *and*:
  - o are receiving intravenous fluids or
  - o are receiving a vasopressor or inotrope

Acute Hospital: A hospital admitting acutely unwell patients – i.e. patients who have a recent onset or exacerbation of a somatic condition and require timely care. Acute hospitals can be owned and run by the government or by a private or other organisation. Hospitals that only admit chronically unwell patients, or only patients for rehabilitation, or only patients for elective surgery are not regarded as acute hospitals and are not eligible for participation in ACIOS. Hospitals, units and wards exclusively for patients with psychiatric conditions are not regarded as acute hospitals.

*In-hospital mortality (co-primary outcome):* Death in-hospital. Patients discharged alive are not followed-up at home.

*1-day and 7-day outcomes:* The defined time for the outcomes is from the point of inclusion of the patient into the study to hospital discharge or death, censored at 7-days.

# 9. Data Handling and Management

The papers containing identifiable patient data for the follow-up of clinical outcomes will be stored within a locked office in each hospital or institution. Data will then be pseudo-anonymised by generation of a unique numeric code and transcribed by local investigators onto an internet based electronic case-record file (e-CRF).

Each patient will only be identified on the e-CRF by their numeric code; thus the central co-ordinating study team cannot trace data back to an individual patient. A participant list will be used in each hospital/site to match identifier codes in the database to individual patients in order to record clinical outcomes and supply any missing data points. This participant list will be stored on a password-protected computer. Access to the data entry system will be based on the principle of least privilege and







will be protected by username and password delivered during the registration process for individual local investigators.

All electronic data transfer between participating hospitals and the co-ordinating institution will be encrypted using a secure protocol (HTTPS/SSL 3.0 or better). Data will be anonymised during the transcription process using the Research Electronic Data Capture (REDCap) tools hosted by Safe Surgery South Africa (SSSA) who will act as the data custodian. REDCap is a secure, web-based application designed to support databases and data capturing for research studies. Soft limits will be set for data entry, prompting investigators when data were entered outside these limits. In countries with poor internet access, paper case record forms may be forwarded to SSSA, for entry by SSSA. Pseudo-anonymised (coded) data may also be sent by encrypted e-mail to the coordinating institution if necessary. Each institution will maintain a secure trial file including a protocol, local investigator delegation log, ethics approval documentation, the participant list, etc. Copies of the relevant protocols, approvals and investigator lists will also be kept securely in an internal drive by SSSA. A final summary of included patients with aggregated data of patients, and outcomes will be produced for each hospital together with final data submission to double check for completeness and accuracy.

Individual patient data provided by participating hospitals remain the property of the respective institution, once the ACIOS report has been published. Once each local co-ordinator has confirmed the data provided from their hospital are both complete and accurate, they will be provided with a spreadsheet of the raw (un-cleaned) data for their hospital. In the ACIOS report, only summary data will be presented publicly, and all national, institutional and patient level data will be strictly anonymised.

## **10.Statistical Analysis**

### 10.1 Sample size calculation

Our plan is to recruit as many hospitals as possible in as many African countries as possible. All eligible patients will be included in each hospital. We do not have a specific sample size.

## 10.2 Statistical analysis

An ACIOS statistical analysis plan (SAP) will be written prior to inspection of the final dataset. Data will be presented at a continental African level. All institutional and national level data will be anonymised prior to publication. Categorical variables will be described as proportions and will be compared using








chi-square tests. Continuous variables will be described as mean and standard deviation if normally distributed, or median and inter-quartile range if not normally distributed. Comparisons of continuous variables between groups will be performed using t-tests, one-way ANOVA or equivalent non-parametric tests as appropriate. Univariate and hierarchical, multivariable, multi-level logistic regression models will be constructed to determine the relationship between the presence of critical illness and mortality and the relationship between essential emergency and critical care provision and mortality.

Results of logistic regression will be reported with 95% confidence intervals. The models will be assessed with predefined sensitivity analyses to explore possible interacting factors and examine any effect on the results. A single final analysis is planned at the end of the study.

#### 11. Ethical Considerations

The study will be carried out in accordance with the ethical principles in the International Conference on Harmonisation and Good Clinical Practice. Ethical approval will be obtained from the University of Cape Town with additional approvals in each country as required by national ethical committees, and from each institution as required by local regulatory requirements. Country Coordinators will be responsible for clarifying the need for ethical and regulatory approvals and for ensuring these are in place prior to data collection. Participating hospitals will not be permitted to record data without providing confirmation that the necessary ethical and regulatory approvals are in place.

The requirement for patient consent may vary according to national regulations. We anticipate that patient consent will not be required by most, or even all, nations on the basis that the study is, in effect, a large-scale clinical audit, the dataset will only include variables documented as part of routine clinical care, and identifiable patient data will not leave the treating hospital. Most importantly, critically ill patients are frequently unable to consent for themselves due to a decreased level of consciousness and a requirement of consent would exclude the very patients we most wish to help. Therefore, we will use 'broadcasting' signage informing patients and families that the site is participating in the study, if required by regulations to ensure patients are aware of the study (Appendix 1). A precedent for this approach was set internationally with the EuSOS and ASOS studies. In EuSOS, consent was waived in 27 of the 28 European countries participating,<sup>37</sup> and in the ASOS-1<sup>38</sup> and ASOS-2<sup>39</sup> consent was waived in the majority of hospitals.








There is an ethical consideration when the study team observes a patient that is critically ill (see the Definitions section 8) requiring urgent care. On these occasions, the study team will immediately notify the clinical team about the patient's condition and provide them with the patient's vital signs. The treating clinicians will therefore be timeously alerted to the status of the patient, and will be able to manage the patient according to local protocols. In each hospital, the study team will offer to document the patients' vital signs in the medical records – as in some low resource hospitals, patients' vital signs are not checked daily due to a lack of human or material capacity, so the project may contribute to an improvement to the standard of care.

As the data will only be submitted once the e-CRFs are complete, and the steering committee will only analyse the data after data collection is complete (and not in real time), the investigators will be unable to intervene in the clinical management of patients.

# 12. Safety considerations

There are no safety considerations relating to the study. There is no risk of harm to either patients or investigators.

# 13. Monitoring and Auditing

ACIOS study documents may be selected by the Sponsor to ensure study activities are conducted according to the protocol, the Sponsor's standard operating procedures, Good Clinical Practice and the applicable regulatory requirements. In participating hospitals, local study documents may also be selected for audit on a local basis. The ACIOS study team will not routinely monitor data collection in individual hospitals or conduct source data verification.

## **14.Study Committees**

## 14.1 Study Management Team

ACIOS will be led by the Study Management Team who will be responsible for study administration, communication between project partners, data collection and data management.








# **14.2 Steering Committee**

A Steering Committee will be responsible for overseeing the study and its scientific conduct.

#### **14.3 Country Coordinators**

Country Co-ordinators will be selected to lead the project within their country and:

- Identify hospitals and local co-ordinators in participating hospitals.
- Assist with translation of study paperwork as required.
- Ensure distribution of research manuals, data collection forms and other materials.
- Ensure necessary regulatory approvals are in place prior to the start date.
- Ensure good communication with the participating sites in the country.

#### 14.3 Local Coordinators

Local co-ordinators in individual hospitals will have the following responsibilities:

- Provide leadership for the study in their hospital.
- Ensure all relevant regulatory approvals are in place for their institution.
- Ensure adequate training of all relevant staff prior to data collection.
- Supervise data collection and assist with problem solving.
- Act as guarantor for the integrity and quality of data collected.
- Ensure timely completion of e-CRFs.
- Communicate with the relevant national coordinator.

#### 15. Dissemination and Publication Plan

The Steering Committee will appoint a writing committee to draft the ACIOS scientific report(s) which will be disseminated in a timely manner. The African Partnership for Perioperative and Critical Care Research (APPRISE) group authorship guidelines will be followed. It is anticipated that a number of secondary analyses will be performed. ACIOS investigators and coordinators will be given priority to lead such analyses and are encouraged to do so. Participation and authorship opportunities will be based on contribution to the primary study. The Steering Committee will consider the quality and validity of any proposed study, the statistical analysis plan, a data sharing agreement, objectives that are in-line with the wider aims of the ACIOS project, scientific validity and the possible effect on the anonymity of participating hospitals prior to granting any requests for additional studies. Where







necessary, a prior written agreement will set out the terms of such collaborations. The Steering Committee must approve the final version of all manuscripts including ACIOS data prior to submission, whether they relate to part or all of the ACOIS dataset. In the event of disagreement within the Steering Committee, the Chief Investigators will make a ruling. Any analysis incorporating ACIOS data from two or more study sites will be considered a secondary analysis and subject to these rules. The full study report will be submitted to the funder and will also be made accessible via clinicaltrials.gov.

#### 16. Deliverables

The main deliverables will be scientific reports of findings for general and specialty journals, abstracts for presentation to national and international meetings including those of the supporting societies and a final report summarising the overall findings.

# 17. Finance and Funding

The ACIOS study is funded by the NIHR through the Global Health Group on Perioperative and Critical Care grant (NIHR133850). The funders will play no role in study design, conduct, data collection, data analysis, reporting or interpretation of the results.

### 18.References

- 1. Kayambankadzanja RK, Schell CO, Gerdin Wärnberg M, et al. Towards definitions of critical illness and critical care using concept analysis. *BMJ open* 2022; **12**(9): e060972.
- 2. Jenson A, Hansoti B, Rothman R, de Ramirez SS, Lobner K, Wallis L. Reliability and validity of emergency department triage tools in low- and middle-income countries: a systematic review. *European Journal of Emergency Medicine* 2018; **25**(3).
- 3. Kruisselbrink R, Kwizera A, Crowther M, et al. Modified Early Warning Score (MEWS) Identifies Critical Illness among Ward Patients in a Resource Restricted Setting in Kampala, Uganda: A Prospective Observational Study. *PloS one* 2016; **11**(3): e0151408.
- 4. Phua J, Faruq MO, Kulkarni AP, et al. Critical Care Bed Capacity in Asian Countries and Regions. *Critical care medicine* 2020.
- 5. Maharaj R, Raffaele I, Wendon J. Rapid response systems: a systematic review and meta-analysis. *Critical care (London, England)* 2015; **19**(1): 254.
- 6. Kayambankadzanja RK, Likaka A, Mndolo SK, Chatsika GS, Umar E, Baker T. Emergency and critical care services in Malawi: Findings from a nationwide survey of health facilities. *Malawi Medical Journal* 2020; **32**(1): 259-63.
- 7. Baker T, Lugazia E, Eriksen J, Mwafongo V, Irestedt L, Konrad D. Emergency and critical care services in Tanzania: a survey of ten hospitals. *BMC health services research* 2013; **13**: 140.








- 8. Kayambankadzanja RK, Schell CO, Mbingwani I, Mndolo SK, Castegren M, Baker T. Unmet need of essential treatments for critical illness in Malawi. *PloS one* 2021; **16**(9): e0256361.
- 9. Schell CO, Gerdin Wärnberg M, Hvarfner A, et al. The global need for essential emergency and critical care. *Critical Care* 2018; **22**(1): 284.
- 10. Schell CO, Khalid K, Wharton-Smith A, et al. Essential Emergency and Critical Care: a consensus among global clinical experts. *BMJ Global Health* 2021; **6**(9): e006585.
- 11. Crawford AM, Shiferaw AA, Ntambwe P, et al. Global critical care: a call to action. *Critical Care* 2023; **27**(1): 28.
- 12. Mekontso Dessap A, Richard J-CM, Baker T, Godard A, Carteaux G. Technical Innovation in Critical Care in a World of Constraints: Lessons from the COVID-19 Pandemic. *American journal of respiratory and critical care medicine* 2023.
- 13. Buowari DY, Owoo C, Gupta L, Schell CO, Baker T. Essential Emergency and Critical Care: A Priority for Health Systems Globally. *Critical care clinics* 2022; **38**(4): 639-56.
- 14. Rudd KE, Johnson SC, Agesa KM, et al. Global, regional, and national sepsis incidence and mortality, 1990–2017: analysis for the Global Burden of Disease Study. *The Lancet* 2020; **395**(10219): 200-11.
- 15. Haagsma JA, Graetz N, Bolliger I, et al. The global burden of injury: incidence, mortality, disability-adjusted life years and time trends from the Global Burden of Disease study 2013. *Injury Prevention* 2016; **22**(1): 3.
- 16. Meara JG, Leather AJ, Hagander L, et al. Global Surgery 2030: evidence and solutions for achieving health, welfare, and economic development. *Lancet* 2015; **386**(9993): 569-624.
- 17. Schell CO, Baker T, al. e. The burden of critical illness among adults in a Swedish region a population-based point-prevalence study; 2023.
- 18. Mboya EA, Baker T, al. e. Critical illness at the Emergency Department of a Tanzanian National Hospital in a three- year period 2019-2021. 13 January 2023, PREPRINT (Version 1) available at Research Square https://doiorg/1021203/rs3rs-2446335/v1.
- 19. Murthy S, Wunsch H. Clinical review: International comparisons in critical care lessons learned. *Critical care (London, England)* 2012; **16**(2): 218.
- 20. Adhikari NK, Fowler RA, Bhagwanjee S, Rubenfeld GD. Critical care and the global burden of critical illness in adults. *Lancet* 2010; **376**(9749): 1339-46.
- 21. Kayambankadzanja RK, Schell CO, Namboya F, et al. The Prevalence and Outcomes of Sepsis in Adult Patients in Two Hospitals in Malawi. *The American journal of tropical medicine and hygiene* 2020.
- 22. Biccard BM, Gopalan PD, Miller M, et al. Patient care and clinical outcomes for patients with COVID-19 infection admitted to African high-care or intensive care units (ACCCOS): a multicentre, prospective, observational cohort study. *The Lancet* 2021; **397**(10288): 1885-94.
- 23. Ilori IU, Kalu QN. Intensive care admissions and outcome at the University of Calabar Teaching Hospital, Nigeria. *Journal of critical care* 2012; **27**(1): 105 e1-4.
- Towey RM, Ojara S. Practice of intensive care in rural Africa: an assessment of data from Northern Uganda. *African health sciences* 2008; **8**(1): 61-4.
- 25. Gombar S, Ahuja V, Jafra A. A retrospective analysis of obstetric patient's outcome in intensive care unit of a tertiary care center. *Journal of anaesthesiology, clinical pharmacology* 2014; **30**(4): 502-7.
- 26. Subbe CP, Kruger M, Rutherford P, Gemmel L. Validation of a modified Early Warning Score in medical admissions. *QJM : monthly journal of the Association of Physicians* 2001; **94**(10): 521-6.
- 27. Kause J, Smith G, Prytherch D, Parr M, Flabouris A, Hillman K. A comparison of antecedents to cardiac arrests, deaths and emergency intensive care admissions in Australia and New Zealand, and the United Kingdom--the ACADEMIA study. *Resuscitation* 2004; **62**(3): 275-82.
- 28. Smith AF, Wood J. Can some in-hospital cardio-respiratory arrests be prevented? A prospective survey. *Resuscitation* 1998; **37**(3): 133-7.
- 29. Kellett J, Deane B. The Simple Clinical Score predicts mortality for 30 days after admission to an acute medical unit. *QJM-An Int J Med* 2006; **99**(11): 771-81.
- 30. Baker T, Blixt J, Lugazia E, et al. Single Deranged Physiologic Parameters Are Associated With Mortality in a Low-Income Country. *Critical care medicine* 2015; **43**(10): 2171-9.







- 31. Baker T, Gerdin M. The clinical usefulness of prognostic prediction models in critical illness. *European journal of internal medicine* 2017.
- 32. Global patient outcomes after elective surgery: prospective cohort study in 27 low-, middle- and high-income countries. *Br J Anaesth* 2016; **117**(5): 601-9.
- 33. Pearse RM, Moreno RP, Bauer P, et al. Mortality after surgery in Europe: a 7 day cohort study. *The Lancet* 2012; **380**(9847): 1059-65.
- 34. Biccard BM, Madiba TE, Kluyts H-L, et al. Perioperative patient outcomes in the African Surgical Outcomes Study: a 7-day prospective observational cohort study. *The Lancet* 2018.
- 35. Baker T, Schell CO, Lugazia E, et al. Vital Signs Directed Therapy: Improving Care in an Intensive Care Unit in a Low-Income Country. *PloS one* 2015; **10**(12): e0144801.
- 36. Bell MB, Konrad D, Granath F, Ekbom A, Martling CR. Prevalence and sensitivity of MET-criteria in a Scandinavian University Hospital. *Resuscitation* 2006; **70**(1): 66-73.
- 37. Pearse RM, Moreno RP, Bauer P, et al. Mortality after surgery in Europe: a 7 day cohort study. *Lancet* 2012; **380**(9847): 1059-65.
- 38. Biccard BM, Madiba TE, Kluyts HL, et al. Perioperative patient outcomes in the African Surgical Outcomes Study: a 7-day prospective observational cohort study. *Lancet* 2018; **391**(10130): 1589-98.
- 39. Biccard BM, du Toit L, Lesosky M, et al. Enhanced postoperative surveillance versus standard of care to reduce mortality among adult surgical patients in Africa (ASOS-2): a cluster-randomised controlled trial. *The Lancet Global Health* 2021; **9**(10): e1391-e401.







# **Appendices**

Appendix 1 – Broadcasting document

| IMPORTANT PATIENT INFORMATION |
|---|
| A research study is being conducted atHospital. |
| The research study is being done by Dr from the Department of |
| Why is this research study being done? |
| To understand how sick patients are in hospital. |
| Why are we telling you about this research study? |
| All patients in this hospital are part of the research study. It is a requirement that some details pertaining to your clinical care are entered into a research study folder. Information from this folder will be used anonymously to understand how sick patients are in hospital, and what we might be able to do to improve the care for sick patients. |
| Will this research study affect my care while I am in hospital? |
| No. You will still receive the same care while you are in hospital. |
| Will my name or any personal details be kept by this research study? |
| No. Your name and personal details will not be kept as part of this research study. All information from the notes will be kept strictly confidential. |
| Are there any risks or benefits associated with this project? |
| No. There are no risks or direct benefits associated with this research study. |
| Who should I contact if I have any questions or concerns? |
| Please contact Dr on telephone |
| If you have questions about your rights or welfare as a participant, please contact the UCT Faculty of Health Sciences Human Research Ethics Committee on +27 (0)21 406 6338. <b>2</b> |







# Appendix 2 – Case record forms (CRFs)

2a: Hospital level CRF

# African Critical Illness Outcomes Study (ACIOS) - Hospital CRF

# **Section 1: Hospital characteristics**

| 1. | Language preference: | ☐ English ☐ F | rench [ | Arabic 🗌 Po | rtuguese 🗌 | Other | |
|---|---|---|---|---|---|---|---|
| 2. | Hospital name: | | ••••• | | | | |
| 3. | Country: | | ••••• | | | | |
| 4. | Level of hospital: | | | | | | |
| | First-level (e.g. district) | Second-level | (e.g. Reg | iional) 🗌 Thi | rd-level (e.g. | University/Central/N | National) |
| 5. | Type of hospital: | Government | | ☐ Private | | ☐ Charitable | |
| 6. | Total number of hospital I | oeds: | Total | | | | |
| 7. | Number of beds in High C | Care Units: | Total | | | | |
| 8. | Number of beds in ICUs: | | Total | | | | |
| 9. | Population served (catchn | nent) of the hospit | tal: | | | | |







# **Section 2: Available Resources**

Are the following available in your hospital?

| | EQUIPMENT | Always | Sometimes | Never | Don' tknow |
|---|---|---|---|---|---|
| 1 | Clock with second hand | 0 | 0 | 0 | 0 |
| 2 | Pulse oximeter & probe | 0 | 0 | 0 | 0 |
| 3 | Blood pressure measuring equipment (eg. sphygmomanometer with a stethoscope) | 0 | 0 | 0 | 0 |
| 4 | Blood pressure cuffs of different paediatric and adult sizes | 0 | 0 | 0 | 0 |
| 5 | Light source (lamp or flashlight) | 0 | 0 | 0 | 0 |
| 6 | Thermometer | 0 | 0 | 0 | 0 |
| 7 | Suction machine (electric or manual) | 0 | 0 | 0 | 0 |
| 8 | Oxygen supply 24h/day<br>(cylinder, concentrator (with<br>electricity supply) or piped<br>oxygen) | 0 | 0 | 0 | 0 |
| 9 | Flow meter (if using cylinder or piped oxygen) | 0 | 0 | 0 | 0 |
| 10 | Leak-free connectors from oxygen source to tubing | 0 | 0 | 0 | 0 |
| 11 | Bag Valve Mask (resuscitator) – neonatal, paediatric and adult sizes | 0 | 0 | 0 | 0 |

| 12 | Sharps disposal container | 0 | 0 | 0 | 0 |
|----|---------------------------|---|---|---|---|
| 13 | External heat source | 0 | 0 | 0 | 0 |

| | CONSUMABLES | Always | Sometimes | Never | Don' tknow |
|---|---|---|---|---|---|
| 14 | Soap or hand disinfectant | 0 | 0 | 0 | 0 |
| 15 | Examination gloves | 0 | 0 | 0 | 0 |
| 16 | Suction catheters of paediatric and adult sizes | 0 | 0 | 0 | 0 |
| 17 | Guedel airways of paediatric and adult sizes | 0 | 0 | 0 | 0 |
| 18 | Pillows | 0 | 0 | 0 | 0 |
| 19 | Oxygen tubing | 0 | 0 | 0 | 0 |
| 20 | Oxygen nasal prongs | 0 | 0 | 0 | 0 |
| 21 | Oxygen face masks of paediatric and adult sizes | 0 | 0 | 0 | 0 |
| 22 | Oxygen face masks with reservoir bags of paediatric and adult sizes | 0 | 0 | 0 | 0 |
| 23 | Masks for Bag Valve Mask<br>(resuscitator) – neonatal, paediatric and<br>adult sizes | 0 | 0 | 0 | 0 |
| 24 | Compression bandages | 0 | 0 | 0 | 0 |
| 25 | Plasters or tape | 0 | 0 | 0 | 0 |







| 26 | Gauze | | | | О | 0 | 42 | fluids (eg. normal saline or<br>Ringer's Lactate) | | 0 | 0 | 0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 27 | Intravenous cannulas of paediatric and adult sizes | C | | ) ( | Э | 0 | | | | | | |
| 28 | Intravenous giving sets | C | ) ( | ) ( | Э | 0 | 43 | 43 Intravenous dextrose fluid (eg. 5%, 10% or 50%) | | 0 | 0 | 0 |
| 29 | Skin disinfectant for cannulation | C | ) ( | ) ( | Э | 0 | 44 | Oxytocin | 0 | 0 | 0 | 0 |
| 30 | Syringes | | | | О | 0 | 45 | Adrenaline | 0 | 0 | 0 | 0 |
| 31 | Nutrition | C | ) ( | ) ( | Э | 0 | 46 | Appropriate antibiotics | 0 | 0 | 0 | 0 |
| 32 | Nasogastric tubes | C | ) ( | ) ( | Э | 0 | 47 | Diazepam | 0 | 0 | 0 | 0 |
| 33 | Lubricant for nasogastric tube insertion | C | ) ( | ) ( | Э | 0 | 48 | Magnesium sulphate | 0 | 0 | 0 | 0 |
| 34 | Intramuscular needles | C | ) ( | ) ( | Э | 0 | 49 | Paracetamol | 0 | 0 | 0 | 0 |
| 35 | Intraosseous cannulas of different sizes | C | ) ( | ) ( | 5 | 0 | 50 | Local anaesthetic (eg. 2% lignocaine) (eg. for intraosseous cannulation) | 0 | 0 | 0 | 0 |
| 36 | Blankets | C | | ) ( | Э | 0 | | | ] | ] | ] | |
| 37 | Facemasks for Infection Prevention and Control | C | | ) ( | 5 | 0 | | | | es | | ow |
| 38 | Aprons or gowns | C | ) ( | ) ( | <b>)</b> | 0 | | HR | Always | Sometimes | Never | Don' tknow |
| 39 | Charts/notes for documentation | C | | ) ( | Э | 0 | 51 | Health workers (eg nurses) with the ability to identify critical illness 24h/day | 0 | 0 | 0 | 0 |
| 40 | Pens | C | ) ( | ) ( | Э | 0 | | | | | | |
| | | | nes | | | wou | 52 | Health workers with the (eg nurses) ability to care for critically ill patients 24hrs/day | 0 | 0 | 0 | 0 |
| | DRUGS | Always | Sometimes | Never | | Don't know | 53 | Senior health worker (eg doctor) who can be called to assist with the care of | 0 | 0 | 0 | 0 |
| 41 | Oral rehydration solution | 0 | 0 | 0 | ) | 0 | | critically ill patients | | | | |

24hrs/day



other care including the definitive care of the underlying





| | TRAINING | Always | Sometimes | Never | Don' tknow | condition (eg. use specific guidelines) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 54 | The health workers are trained in the identification of critical illness | 0 | 0 | 0 | 0 | GUIDEL | INES | Always | Sometimes | Never | Don' tknow |
| 55 | The health workers are trained in the care of critically ill patients | 0 | 0 | 0 | 0 | 61 There are writt guidelines for t identification o illness | he | 0 | 0 | 0 | 0 |
| | | | | | | 62 There are writt guidelines for t care of critically | he essential | 0 | 0 | 0 | 0 |
| | ROUTINES | Always | Sometimes | Never | Don' tknow | INFRASTRU | INFRASTRUCTURE | | Sometimes | Never | Don' tknow |
| 56 | The hospital has well-<br>defined routines for the<br>identification of critical<br>illness | 0 | 0 | 0 | 0 | 63 Designated tria (area for the id of critical illnes | ge area<br>entification | Always | Some | ž | Don' |
| 57 | The hospital has well-<br>defined routines for<br>managing critically ill<br>patients | 0 | 0 | 0 | 0 | Out-Patient De<br>or Emergency U<br>the hospital wh<br>patients arrive) | partment<br>Unit (area of<br>nere | 0 | 0 | 0 | 0 |
| 58 | There is a routine for the provision of EECC without | | | | | 64 Running water | | 0 | 0 | 0 | 0 |
| | taking into account patients' ability to pay | 0 | 0 | 0 | 0 | 65 Designated spa<br>care of critically<br>(eg. a bay, ward | y ill patients | 0 | 0 | 0 | 0 |
| 59 | There are routines for who<br>and how to call to seek<br>senior help 24hrs/day, 7<br>days/week | 0 | 0 | 0 | 0 | unit) 66 Areas for separ managing patie | ents with a | | | | |
| 60 | There are routines for integrating EECC with | 0 | 0 | 0 | 0 | suspected or co<br>contagious dise<br>those without | | 0 | 0 | 0 | 0 |







2b: Patient's bedside CRF







# African Critical Illness Outcomes Study (ACIOS) – Patient CRF

| Clinical assessment | |
|---|---|
| Date of assessment: d d m m y y y y | |
| Vital signs done by the investigating team: Y N If no, specify Vital signs from patient records Not d | one |
| Position of patient: | |
| ☐ Lying flat on back(<30°) ☐ Lying on side ☐ Head-up(30°-60°) ☐ Sitting(>60°) ☐ Head-down ☐ Otl | her |
| Airway patency: | |
| Conscious level (AVPU): Alert Responds to Voice Responds to Pain Unresponsive | |
| Heart rate /min Oxygen saturation % Respiratory rate /min | |
| Systolic blood pressure /mmHg Diastolic blood pressure /mmHg | |
| Currently receiving IV fluids Y N Receiving oxygen (now) Y I | N |
| Receiving vasopressor/inotrope (now) | N |
| Circle the worst pain you had in the last 24 hours: 0 (no pain) 1 2 3 4 5 6 7 8 9 10 (worst pain you can image | ine) |
| Other information | |
| Date of hospital admission: d m m y y y Urgency of admission: Emergency/acute Elect | ive |
| Age years Sex M F | |
| Ward type: Medical Surgical Maternal Other | |
| Ward level: General ward High care unit/HDU ICU | |
| Main category for admission: Non-communicable disease Maternal health Trauma Infection | n |
| Known chronic disease or pregnancy (tick all that apply): | |
| Pregnant Hypertension Diabetes Cancer COPD / Asthma | |
| ☐ Heart Disease ☐ HIV / AIDS ☐ Tuberculosis ☐ Other ☐ None | |
| Any surgery during this admission: $\square$ Y $\square$ N Treatment limitations (e.g. not for resuscitation): $\square$ Y $\square$ | ] N |
| Follow-up | |
| Total days in hospital from admission to discharge | |
| Status at 7 <sup>th</sup> day in-hospital after clinical assessment: Discharged Alive Alive still in-hospital Died | k |
| Date of discharge or death d d m m y y y y | |
| ACIOS unique patient ID | |
| \$ | |
| Patient name: DOB d d m m y y y y | |
| Patient hospital number Ward Bed | |













#### **Definitions:**

Position of patient: The position the patient is in the bed/chair when the investigating team arrive at the bedside. The number of degrees refers to the angle of the head and body compared to the legs.

**Airway patency:** Normal is an unobstructed airway. Partial obstruction may be indicated by stridor, secretions in the airway identified by gurgling, or snoring. Complete obstruction is evident by a see-saw chest movement (chest down and abdomen up with attempted breathing against a closed glottis). Complete obstruction is an airway emergency and requires calling the attending clinical team immediately.

Conscious level AVPU: Measurement of conscious level. Is the patient Alert = A. If they are not alert but they respond to your voice = V. If they don't respond to voice but respond to a painful stimulus = P. If they remain unresponsive even with a painful stimulus = U (unresponsive).

Currently receiving IV fluids: At the time of clinical assessment, the patient is receiving IV fluids if IV fluids are hanging at the bedside, and currently dripping into an intravenous cannula, or the patient has been receiving fluids as described within the previous few minutes but is now finished and a new fluid is being prepared to be administered.

Receiving oxygen (now): At the time of clinical assessment, the patient is receiving oxygen if supplementary oxygen is currently flowing into a nasal cannula, face mask or other delivery device that is correctly fitted so that oxygen is entering the patient's lungs.

Receiving vasopressor/inotrope (now): Ongoing care with a vasopressor or inotrope infusion – for example noradrenaline, adrenaline, dopamine or dobutamine.

Airway action (now): An action to open the airway or maintain a free airway. For example: chin lift, jaw thrust, oro-pharyngeal airway, naso-pharyngeal airway, intubated patient.

High care unit/HDU: A unit or ward or part of a ward which is dedicated to providing an increased level of care when compared to a general ward. High care units often have increased nurse:patient ratios, more equipment and more advanced care such as oxygen, CPAP, vasopressors etc. This does *not* include units with mechanical ventilation, as that is an ICU. Includes recovery rooms providing an increased level of care.

ICU: A unit or ward which is dedicated to providing an increased level of care when compared to a general ward or high care unit including mechanical ventilation

Main category for admission: The main diagnosis or reason that the patient is being treated in hospital.

Treatment limitations: A patient has a treatment limitation if the clinical team have made the clinical judgement that some treatments would not be in the patient's best interest. For example "DNR" (do not resuscitate in the event of a cardiac arrest), or "Not for ICU" in the event of deterioration.

Days in hospital: Total number of days in hospital from admission.

Status at hospital discharge or 7th day in-hospital after clinical assessment: The survival status of the patient at hospital discharge, or at the 7th day after clinical assessment (if the patient had not yet been discharged). The study is censored at the 7th day after clinical assessment.

#### Guidance for use of paper case record form (CRF)

- Investigators should write the patient's name and date of birth on the bottom of the CRF. When you
  enter the data on the internet based CRF you will receive an ACIOS patient ID. Please write this on the
  paper CRF as well in case we need to contact you to check your data.
- The clinical assessment and the patient's vital signs MUST be completed at the same time by the investigating team. Only in exceptional circumstances can the vital signs data be taken from the medical records.
- Please take care to enter the date clearly and correctly. Mistakes are common data describing time and date.